CLINICAL TRIAL: NCT04155021
Title: Knowledge and Attitude in Perioperative Erythrocyte Transfusion in Medical Personnel of the Department of Anesthesiology and Department of Orthopedic Surgery in Siriraj Hospital
Brief Title: Knowledge and Attitude in Perioperative Erythrocyte Transfusion in Medical Personnel in Siriraj Hospital
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Assoc Prof, Siriraj Hospital
Other Study IDs: SIRB421
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Transfusion-dependent Anemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to explore the correlation between knowledge and attitude in perioperative erythrocyte transfusion in medical personnel.

DETAILED DESCRIPTION:
Inappropriate erythrocyte transfusion is still have high incidence even lots of the transfusion guidelines and researches was launched. Unnecessary or delayed transfusion can cause morbidity and mortality. This study is descriptive research, questionnaire based survey conducted to explore the correlation between knowledge and attitude in perioperative erythrocyte transfusion in medical personnel in Siriraj Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Post-graduated medical personnel in Siriraj Hospital

Exclusion Criteria:

* Post-graduated medical personnel in Siriraj Hospital who refuse to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Post-graduated medical personnel in Siriraj Hospital who associated with erythrocyte transfusion practice.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Knowledge in perioperative erythocyte transfusion in medical personnel in Siriraj Hospital | 10 minutes
  We aim to explore the reason of high incidence of inappropriate transfusion by conduct the questionnaire, about knowledge and attitude in perioperative erythocyte transfusion in medical personnel in Siriraj Hospital. Knowledge part will measure followed by transfusion guideline of Hematology and Anesthesiology, Siriraj Hospital and attitude toward perioperative transfusion will collect and analyse

SECONDARY OUTCOMES:
Attitude in perioperative erythocyte transfusion in medical personnel in Siriraj Hospital | 10 minutes
  We aim to explore the reason of high incidence of inappropriate transfusion by conduct the questionnaire, about knowledge and attitude in perioperative erythocyte transfusion in medical personnel in Siriraj Hospital. Knowledge part will measure followed by transfusion guideline of Hematology and Anesthesiology, Siriraj Hospital and attitude toward perioperative transfusion will collect and analyse

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand